CLINICAL TRIAL: NCT06288776
Title: Clinical Efficacy of Azadirachta Indica Based Herbal Mouthwash in Treating the Hypersensitivity of Teeth
Brief Title: Efficacy of Azadirachta Indica Based Herbal Mouthwash in Treating the Tooth Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Afsheen Mansoor, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOD/ERB/2023/22-04
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Tooth Sensitivity
Keywords: Azadirachta indica; Gingival Index; Herbal; Mouthwash; Tooth sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: In this study, participants will be selected by consecutive non-random sampling technique.
Masking Description: Single-blinded study where participant will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Group (Experimental): Participants will be assessed for their tooth sensitivity (VAS scoring) and after giving herbal based mouthwash sensitivity will be assessed after 3 months
  Interventions: Diagnostic Test: Herbal based mouthwash

INTERVENTIONS:
Diagnostic Test: Herbal based mouthwash — Herbal based mouthwash will be used to treat the tooth sensitivity in participants having VAS score values of tooth sensitivity ranging between 30-80

SUMMARY:
Type of study: Single-blinded clinical trial to evaluate the effectiveness of Azadirachta indica based Herbal mouthwash to treat the tooth sensitivity in patients.

Participants aged 20 years and above having Gingival Index score 3 will be included in the study. Their tooth sensitivity will be checked initially and then they will be given Herbal based mouthwash for 3 months. Again, their tooth sensitivity shall be checked after 3 months.

DETAILED DESCRIPTION:
In this study Herbal based mouthwash will be evaluated for eliminating the tooth sensitivity in the participants having Gingival Index score 3 with VAS scores for sensitivity ranging between 30-80 . Consecutive non-random sampling technique will be used in this study where Participants included will be assessed for tooth sensitivity through Visual Analogue Scale (VAS) initially for base line readings. These participants will be given Azadirachta indica based Herbal mouthwash for three months and then again their tooth sensitivity will be assessed by Visual Analogue Scale (VAS) for final readings. The mean values of VAS scoring both before and after the usage of herbal mouth wash will be compared to investigate the clinical efficacy of this mouthwash in treating the tooth sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good general health and no allergy
* Patients who have not used any mouthwash in last 3 month
* Study teeth shall be free of decay and restoration
* Study teeth shalll not be mobile
* Study teeth shall have the Gingival Index score 3
* Participants shall be able to read ,write and willing to give consent.

Exclusion Criteria:

* Patients with poor general health and allergies
* Patients who have used any mouthwash in last 3 months
* Teeth with decay and restorations
* Teeth with mobility
* Teeth with Gingival Index score more than 3
* Participants that wonn't be able to read ,write and willing to give consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Toothsensitivity declination with herbal based mouthwash | 3 months
  Evaluation of herbal based mouth wash in eliminating the tooth sensitivity ranging between VAS scores 30-80.

CONTACTS AND LOCATIONS:
Overall Officials: Afsheen Mansoor, PhD, Principal Investigator — School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad.
Locations (1):
- Afsheen Mansoor, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall C, Sufi F, Milleman JL, Milleman KR. Efficacy of a 3% potassium nitrate mouthrinse for the relief of dentinal hypersensitivity: An 8-week randomized controlled study. J Am Dent Assoc. 2019 Mar;150(3):204-212. doi: 10.1016/j.adaj.2018.10.023. PMID 30803493